CLINICAL TRIAL: NCT05136157
Title: Intravenous Bolus-infusion Versus Sliding Scale of Insulin for Intra-operative Glycemic Control in Elective Laparotomy Surgeries
Brief Title: Intravenous Bolus-infusion Versus Sliding Scale of Insulin for Intra-operative Glycemic Control
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ghada M.Samir, Assistant Professor of Anesthesia, Intensive care and Pain Management, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R 16/2020/2021
Record Dates: First submitted 2021-10-08; First posted 2021-11-29 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Intraoperative Complications
Keywords: Insulin; Intra operative; Sliding scale; Bolus- infusion
MeSH Terms: conditions — Intraoperative Complications; Insulin Resistance | interventions — Insulin, Short-Acting

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Active Comparator): Bolus-Infusion approach of rapidly acting crystalline insulin. The patient intra-operative blood glucose will be divided by 100. The resultant rapidly acting crystalline insulin units will be given intravenously over 10 minutes, and then continued as an intra-venous infusion per hour. The Capillary Blood Glucose (CBG) will be measured every 30 minutes and in the PACU with readjustment of the bolus-infusion dose as required
  Interventions: Drug: Rapid-Acting Insulin
- Control group (Active Comparator): The sliding scale approach of rapidly acting crystalline insulin will be used according to the intra-operative blood glucose; 4 IU of insulin will be given when the CBG 180-250 mg/dl, 6 IU of insulin will be given when the CBG 251-300 mg/dl, 8 IU of insulin will be given when the CBG 301-350 mg/dl and 10 IU of insulin will be given when the CBG 351-400 mg/dl (5). The CBG will be measured every 30 minutes and in the PACU.
  Interventions: Drug: Rapid-Acting Insulin

INTERVENTIONS:
Drug: Rapid-Acting Insulin — 50 IU of rapid acting insulin taken by a 100 units (1ml) insulin syringe will be added to a 50 ml syringe containing normal saline (NS) to have a total volume of 50 ml with a concentration of 1 IU of insulin per 1 ml of NS
  Other Names: Crystalline insulin

SUMMARY:
Pre-operative blood glucose (BG) concentrations in type 2 diabetic patients undergoing elective non-cardiac surgery; have an increased incidence of in-hospital morbidity for cardiopulmonary and infectious complications. Also, hyperglycemia is associated with increased production and impaired scavenging of oxygen reactive species, polymorph nuclear neutrophil dysfunction and decreased intracellular killing, resulting in poor wound healing and increased risk of infection. Thus, perioperative optimal glucose management contributes to reduced morbidity and mortality. Recommendations favor moderate levels of capillary blood glucose (CBG); maintaining it in the range of 140-180 mg/dl.

Peri-operative doses of rapidly acting insulin for glycemic control could be done by the sliding scale or the bolus-infusion approaches. The sliding scale of insulin is commonly used to manage peri-operative hyper-glycaemia. It involves administering prescribed doses of insulin when the CBG is within determined ranges and withholding insulin when the CBG is within normal range. When used as a sole therapy; it results in under-insulinisation and thus hyper-glycaemia. The use of a dynamic insulin regimen like the intravenous bolus-infusion approach; allows adjusting the blood glucose level according to the insulin sensitivity of each patient, thus, better glucose control and less variations than the intermittent intravenous bolus of short-acting insulin in the sliding scale despite the same blood glucose target.

DETAILED DESCRIPTION:
compare the rapidly acting insulin injection via the bolus-infusion approach (Study group) to the sliding scale approach (Control group) as regards the intra-operative glycemic control

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status II patients
* aged 21-65 years
* known to have type1 or 2 diabetes mellitusw
* pre-operative fasting blood glucose level ˂ 350 mg/dl
* scheduled to undergo elective laparotomy surgeries
* expected to exceed 2 hours duration under general anesthesia

Exclusion Criteria:

* Patients' refusal
* diabetic ketoacidosis
* hyperglycemic hyperosmolar syndrome
* serum potassium ˂3.5 mEq/L
* HbA1c >8.5%.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
intra-operative CBG level between 140- 180 mg/dl all over the operation | 7 months
  Base line CBG will be measured for all patients then every 30 minutes and in the PACU

SECONDARY OUTCOMES:
Total IU of rapidly acting insulin given to the patient | 7 months
  total units of insulin given to the patient will be calculated in the PACU
Peri-operative changes in serum potassium | 7 months
  Base line serum potassium will be compared to that measured in the PACU

CONTACTS AND LOCATIONS:
Locations (1):
- Ain-Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No